CLINICAL TRIAL: NCT02844075
Title: A Phase II Trial of Preoperative Chemoradiotherapy and MK-3475 for Esophageal Squamous Cell Carcinoma (ACTS-29)
Brief Title: Preoperative Chemoradiotherapy and MK-3475 for Esophageal Squamous Cell Carcinoma (ACTS-29)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0199
Record Dates: First submitted 2016-07-08; First posted 2016-07-26 (Estimated); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; pembrolizumab; PD-1; neoadjuvant; chemoradiation
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pembrolizumab (Experimental)
  Interventions: Drug: MK-3475(pembrolizumab)

INTERVENTIONS:
Drug: MK-3475(pembrolizumab) — Neo-adjuvant chemoradiation period:The treatment consisted of taxol, carboplatin, pembrolizumab and radiation. The radiation treatment comprises 44.1Gy (2.1Gy/Fr, total 21Fr) and that will be about 5 weeks. Intensity modulated RT (IMRT) or 3D CRT (three-dimensional conformal radiotherapy) will be allowed.
  Surgery:Before surgery, abdomen/chest CT scan, endoscopic ultrasound (EUS), and gastroscopy with biopsy will be done. Surgery should be done within 12 weeks after last neo-adjuvant treatment.
  Adjuvant period:Adjuvant treatment with pembrolizumab 200mg every 2week (maximum 2 years) should be performed within 8 weeks after surgery (recommended period : 3-6 weeks after surgery). Gastroscopy and abdomen/chest CT scan will be performed at 6 month after surgery.

SUMMARY:
In this study, participants with esophageal squamous cell carcinoma will receive preoperative chemoradiotherapy with paclitaxel,carboplatin and pembrolizumab then undergo surgery. The primary study hypothesis is that adding pembrolizumab will increase complete pathologic response rate at surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ESCC
2. Clinical stage T1N1-2 or T2-34aN0-12 (AJCC 7 TNM classification)
3. No evidence of metastasis
4. Be willing and able to provide written informed consent/assent for the trial.
5. Be 20 years of age on day of signing informed consent.
6. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion through repeated biopsies. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    - Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has another malignancy within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative surgery, or in situ cervical cancer.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of, or any evidence of active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
17. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong MH, Shin SK, Choi SJ, Ahn BC, Kim HR, Park SY, Kim DJ, Lee CG, Cho J, Kim JH, Kim HR, Kim YH, Lee GT, Park SR, Lee SK, Cho BC. Preoperative chemoradiotherapy plus pembrolizumab for esophageal squamous cell carcinoma (ACTS-29). Esophagus. 2026 Jan;23(1):99-110. doi: 10.1007/s10388-025-01165-0. Epub 2025 Dec 25. PMID 41449287

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 60 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 28

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response Rate
Description: The primary endpoint of phase II study is to assess complete pathologic response rate. Definition of complete pathologic response is "no cancer cell, including lympho nodes" which corresponds with tumor regression score 0. Definition of pathologic response is as follows. Tumor regression score Grade 0 and 1 will be defined as "responder" and 2 and 3 will be considered as "non-responders"
Time Frame: Up to 3 years
Population: Underwent surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
Participants | 6
Statistical Analysis 1: Comparison: Pembrolizumab; Test type: Superiority; For sample size calculation, Minimax design to evaluate the null hypothesis that the true pCR rate will be 10% and the alternative hypothesis that the pCR rate≥ 30%, with type I error (α) level of 10% and type II error (β) of 0.10. If 1 or more successes are observed in the first 16 patients, accrual for that stratum will be continued until a total of 25 patients. If, of these 25 patients, 5 or more pCR, an additional investigation is warranted. Allowing for a follow-up loss rate of 10 %, the total sample size is expected as 28. For biomarker evaluation, the categorical groups were investigated to evaluated possible association with response and/or survival. Associations were analyzed by χ2 test or Fisher's exact test for categorical variables. The Kaplan-Meier method was used to analyze survival outcomes (EFS, OS, and DFS). To compare PD-L1 expression between paired pre- and post-neoadjuvant treatment with associated of pCR, the Wilcoxon signed-rank test was used

2. Secondary Outcome: Disease Free Survival
Description: Disease free survival is defined from the time of surgery to initial replace or death.
Time Frame: Up to 3 years
Population: Underwent surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
months | 17.9 [0.9 to 27.6]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined from the time of enrollment to death or last follow-up date.
Time Frame: Up to 3 years
Population: Enrollment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
months | 33.6 [23.8 to 36.0]

4. Secondary Outcome: Pathologic Response Rate
Description: Pathologic response rate is defined as tumor regression score. A score of '0' means 'No cancer cell, including lymph nodes'. A score of '1' means 'Single cells or small groups of cancer cells'. A score of '2' means 'Residual cancer cells outgrown by fibrosis'. A score of '3' means 'Minimum or no treatment effect'.
Time Frame: Up to 3 years
Population: Underwent surgery
Measure: Number; unit: participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 26
participants
  Score '0' | 6
  Score '1' | 10
  Score '2' | 10
  Score '3' | 0

5. Secondary Outcome: Safety According to Common Terminology Criteria for Adverse Events (CTCAE) 4.03
Description: Grade 3-4 adverse events occurring during the neoadjuvant period (no death)
Time Frame: Up to 3 years
Population: Enrollment
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
percentage of participants | 25

6. Secondary Outcome: Event Free Survival
Description: Event free survival is defined from the time of enrollment to 'event' included disease recurrence.
Time Frame: Up to 3 years
Population: Enrollment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
months | 11.0 [0.9 to 27.6]

ADVERSE EVENTS:
Time Frame: During Neoadjuvant and Adjuvant Period (Up to 3.0 years) - Received neoadjuvant chemoradiotherapy with pembrolizumab - (Underwent surgery) Adjuvant pembrolizumab
Description: according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/28
Serious Adverse Events (participants affected / at risk) | 10/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=28)
Anorexia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 2
General weakness (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Hypothyroidism (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=28)
Neutropenia (Blood and lymphatic system disorders) | 14
Nausea (Gastrointestinal disorders) | 7
Esophagitis (Gastrointestinal disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 4
Fatigue (General disorders) | 11
General weakness (General disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 9
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 3
Weight loss (Investigations) | 3
Colitis (Gastrointestinal disorders) | 7
Hypothyroidism (Endocrine disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Hepatitis (Hepatobiliary disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT02844075/Prot_SAP_000.pdf